CLINICAL TRIAL: NCT01359007
Title: A Phase II Study Evaluating the Rate of R0 Resection (Microscopically Negative Margins) After Induction Therapy With 5- Fluorouracil, Leucovorin, Oxaliplatin, Irinotecan (FOLFIRINOX) in Patients With Borderline Resectable or Locally Advanced Inoperable Pancreatic Cancer.
Brief Title: FOLFIRINOX in Patients With Inoperable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The principal investigator terminated the study due to inactivity and low enrollment
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1977
Record Dates: First submitted 2011-05-23; First posted 2011-05-24 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Adenocarcinoma of Pancreas
Keywords: Locally advanced unresectable adenocarcinoma of pancreas; Borderline resectable adenocarcinoma of pancreas
MeSH Terms: interventions — Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRINOX (Experimental): Combination of drugs (Irinotecan, Oxaliplatin, Leucovorin, and 5-Fluorouracil (5-FU)) known as FOLFIRINOX every 2 weeks for 4 treatments. At the end of 4 cycles, patients will be re-evaluated for resectability by CT scan within 28 days of the last dose of chemo. If found amendable to surgery, patient will proceed with resection, and type of resection (R0 or R1) will be recorded.
  Interventions: Drug: Irinotecan, Oxaliplatin, Leucovorin, 5-FU

INTERVENTIONS:
Drug: Irinotecan, Oxaliplatin, Leucovorin, 5-FU — 5-FU 2400 mg/m2 IV continuous infusion for 46-48 hours Days 1-3 for 2 weeks 5-FU 400 mg/m2 IV Bolus Day 1 Oxaliplatin 85 mg/m2 IV over 120min +/-30 min. Day 1 Irinotecan 180 mg/m2 IV to run over 90 min +/- 30 min Day 1 Leucovorin (Before bolus 5-FU) 400 mg/m2 IV over 120 min. +/- 30 Day 1 May give oxaliplatin and leucovorin concurrently

SUMMARY:
The prognosis of patients with locally advanced unresectable pancreatic cancer is poor, and the median survival is less than 1 year. FOLFIRINOX therapy, which induces tumor downstaging sufficient to allow surgical resection, could improve the overall survival of patients with locally advanced pancreatic cancer. Based on the FOLFIRINOX regimen for advanced pancreatic cancer, a phase II study of this regimen in patients with locally advanced unresectable and borderline pancreatic cancer is planned to determine the rate of conversion to operability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced unresectable or borderline resectable adenocarcinoma of pancreas
* Patients must have measurable disease as defined by RECIST 1.1 RECIST evaluations must have occurred within 4 weeks prior to study entry
* No evidence of hepatic or pulmonary metastatic disease by CT or CT/PET scans
* Male or non-pregnant and non-lactating female age > or equal to 18 years and < or equal to 70 years of age
* Patient must have received no prior therapy for the treatment of locally advanced unresectable or borderline resectable pancreatic cancer
* Patients must have adequate blood counts at baseline and blood chemistry levels
* Patient has ECOG Performance Status 0 to 1

Exclusion Criteria:

* Patients with islet cell neoplasms excluded
* Patients with known brain metastases
* Therapeutic Coumadin for a history of pulmonary emboli or deep vein thrombosis (DVT)
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Known infection with HIV, hepatitis B or hepatitis C
* Major surgery or vascular device placement within 4 weeks prior to Day 1 of treatment in study
* Prior chemotherapy or radiation for pancreatic cancer
* History of allergy or hypersensitivity to the study drugs
* Patient is enrolled in any other clinical protocol or investigational trial
* Metastatic disease on radiological staging
* Prior malignancy within last 3 years
* Significant cardiac disease
* Any prior gastrointestinal (GI) disease or history of prior pelvic or abdominal radiation in which in opinion of the investigator may place the patient at increased risk
* peripheral sensory neuropathy > or equal to grade 2 at baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Pant, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FOLFIRINOX
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 60 [52 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  sex: Female | 2
  sex: Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 1
  Race: White | 3
  Race: More than one race | 1
  Race: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: To Estimate, Among Patients With Locally Advanced Unresectable and Borderline Resectable Pancreatic Cancer, the Proportion in Whom R0 Resection is Achieved After Neoadjuvant Therapy.
Time Frame: 2 years
Population: Data was not collected from any single study participant.
Groups:
- 5-FU, Leucovorin, Oxaliplatin, Irinotecan: As per above
Arm/Group | 5-FU, Leucovorin, Oxaliplatin, Irinotecan
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Patients Whose Pancreatic Cancer is Operable (Resulting in R0 or R1 Resection) Following Induction Therapy.
Time Frame: 2 years
Population: Data was not collected from any single study participant
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Rate (Either Complete Response (CR) or Partial Response (PR) by RECIST 1.1 Criteria)
Time Frame: 2 years
Population: Data was not collected from any single study participant.
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Time Frame: 2 years
Population: Data was not collected from any single study participant.
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Experienced Toxicity
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | FOLFIRINOX
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX (N=5)
Post-operative bleeding (Injury, poisoning and procedural complications) | 1 (1) — Post-op bleeding following surgical resection
biliary obstruction (Hepatobiliary disorders) | 1 (1) — Biliary obstruction requiring stent

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes